CLINICAL TRIAL: NCT00955045
Title: A Long-Term, Multicenter, Open-Label, Safety Study With a Flexible Dose Range of KW-6002 as Treatment for Parkinson's Disease in Patients With Motor Response Complications on Levodopa/Carbidopa Therapy
Brief Title: A Long-Term, Safety Study With a Flexible Dose Range of KW-6002 in Patients With Motor Response Complications on Levodopa/Carbidopa Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Other Study IDs: 6002-US-007
Record Dates: First submitted 2009-08-04; First posted 2009-08-07 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease
Keywords: long-term tolerability and safety; istradefylline treatment; levodopa/carbidopa
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline

ARMS (1):
- istradefylline (Experimental)
  Interventions: Drug: istradefylline

INTERVENTIONS:
Drug: istradefylline

SUMMARY:
The primary objective of this study was to establish the long-term tolerability and safety of istradefylline treatment in subjects with Parkinson's disease treated with levodopa/carbidopa. In addition, treatment response and maintenance of response were assessed.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects were:

* male or female
* at least 30 years of age
* had completed participation in a prior double-blind istradefylline trial
* met United Kingdom's Parkinson's Disease Society (UKPDS) brain bank criteria (Step 1 and Step 2) for Parkinson's disease and the severity of the Parkinson's disease was defined as Stages 2-4 on the Modified Hoehn and Yahr Scale while in the OFF state
* had been treated with levodopa for at least 1 year
* had been on a stable Parkinson's disease regimen within normal therapeutic ranges including levodopa for at least 4 weeks before Baseline
* were currently taking at least 4 doses of levodopa per day (3 doses per day if at least 2 doses contained slow-release formulation)
* had predictable end-of-dose wearing-off

Exclusion Criteria:

* none

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-08; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- 48 Centers in the US and 4 in Canada, Princeton, New Jersey, United States